CLINICAL TRIAL: NCT06343909
Title: Comparison of Intrinsic Foot Muscle Strengthening and Hip Abductor Strengthening on Pain, Range of Motion, Function, Foot Arches and Knee Alignment in Patients With Knee Osteoarthritis
Brief Title: Foot and Hip Abductor Strengthening in Patients With Knee Osteoarthritis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0197Ayesha
Record Dates: First submitted 2024-03-25; First posted 2024-04-03 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis, KOOS, Strengthening Exercises
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hip abductor strengthening exercise along with conventional exercises (Active Comparator): Hip abductor strengthening Participant was positioned in side lying with bottom leg hip abducting to a 45-degree and knee in flexion. The uppermost leg was actively abducted while it remains in slight extension making sure no rotation occurred. Participant was instructed to hold the leg in that position for 5-10 seconds and then to lower it to resting position.
  Participant was instructed to repeat the exercise with weight cuff attached to the proximal part of ankle
  Interventions: Other: Hip abductor strengthening exercise
- intrinsic foot muscle strengthening exercise along with conventional exercises (Active Comparator): Wring towel with feet:
  . Patient in sitting position, place a hand towel flat on the floor pull the towel towards your heel.
  Grapping object with toes:
  Sitting, place the object flat on the floor.
  . Hold it for a second and then according to the resistance of the release it.
  Toe abduction (hallux and 2nd toe):
  Sitting place a small band between the hallux and second toe. Open and separate your toe and then squeeze the toe against the resistance of elastic. Always leave your feet resting on the floor..
  Toggle toe support:
  Sitting with feet resting on the floor, alternately touch the first and fifth toes on the floor. Be careful not to move your knees.
  Interventions: Other: Intrinsic foot muscle strengthening along with conventional exercises

INTERVENTIONS:
Other: Hip abductor strengthening exercise — in this group 15 participants will perform hip abductor streghtning along with conventional exercises .protocol for 8 weeks 24 sessions (3 sessions in a weak) and 10 sec rest between each segment,3 sets and 10 reputations will be performed.
  Other Names: conventional exercises
  Arms: Hip abductor strengthening exercise along with conventional exercises
Other: Intrinsic foot muscle strengthening along with conventional exercises — in this group 15 participants will perform Intrinsic foot muscle strengthening along with conventional exercises .protocol for 8 weeks 24 sessions (3 sessions in a weak) and 10 sec rest between each segment,3 sets and 10 repitations will be performed.
  Arms: intrinsic foot muscle strengthening exercise along with conventional exercises

SUMMARY:
The study will be Randomized controlled trail, Subject diagnosed with knee osteoarthritis meeting predetermined inclusion and exclusion criteria will be divided into two groups.

Pre assessment will be done using pain, ROM, function, foot arches and knee alignment as subjective measurement through KOOS questionnaire, goniometer, 2D frontal plane projection, Berkemann foot prints using ink and paper ,30s chair stand test, nine step stair climb,40m fast paced walk test,Global rating of change score respectively . One group will be treated with hip abductor strengthening exercise along with conventional exercises and second group will be treated with intrinsic foot muscle strengthening exercise along with conventional exercises. Post treatment values recorded after the session.After data collection from defined study setting,data will be entered and analyzed at Riphah International University,Lahore

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is a leading cause of joint pain1 and disability2 in middle- and older-aged individuals, and is one of the most commonly managed conditions in primary care3. Recent incidence rates suggest around 6% of people aged over 45 years develop knee symptoms. Knee OA symptoms and radiographic change that worsen over time can lead to costly surgical intervention.

Compressive forces on the knee caused by knee adduction moment on the medial compartment of the joint are associated with the severity of the disease and intensity of pain. In addition, decreased strength of the quadriceps is one of the contributing factors for the onset of the disease.

short foot exercises (SFE) have shown to be effective using the IFM and excluding the EFM found that SFE contracted the intrinsic muscles of the foot to increase the inner arch of the foot, thereby shortening the longitudinal arch.Pronated foot is deeply related to the medial longitudinal arch (MLA) where the presence of a pronated foot consequently leads to a decrease in the MLA.

ELIGIBILITY:
Inclusion criteria:

* pain at medial side of the knee.
* patient can walk without walking aids.

Exclusion criteria:

* patient with previous hip, knee and ankle surgery.
* patient who received intraarticular injection.
* patient with neurologic and muscle problem.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-11-23 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Knee Osteoarthritis Outcome Score (KOOS) | 8 weeks
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a questionnaire designed to assess short and long-term patient-relevant outcomes following knee injury.A Likert scale is used and all items have five possible answer options scored from 0 (No problems) to 4 (Extreme problems).
Berkemann foot prints | 8 weeks
  For arch measurement, the longitudinal and horizontal arch lengths were recorded for the left and right feet to create a static standing position using a Berkemann footprint

SECONDARY OUTCOMES:
Frontal plane projection | 8 weeks
  Two-dimensional (2D) frontal-plane projection angles of hip and knee alignment were measured during a single-leg step-down performed from a 15-cm step
Goniometer | 8 weeks
  Universal Goniometer (UG) An instrument called a goniometer is used to measure a joint's range of motion.
30 seconds chair stand test | 8 weeks
  This test used to measure physical function.
Overall self-perception by Global Rating of Change Score | 8 weeks
  Overall self-perception will be evaluated by the Global Rating of Change Score, an 11-point scale designed to quantify a patient's improvement or deterioration over time. Higher scores indicate better recovery from KOA
9 step stairs climb test. | 8 weeks
  This test used to measure physical function.
40-m fast-paced walk test | 8 weeks
  This test used to measure physical function.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Sanaullah, MS, Principal Investigator — Riphah International University
Locations (1):
- THQ hospital KRK., Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Messier SP, Mihalko SL, Beavers DP, Nicklas BJ, DeVita P, Carr JJ, Hunter DJ, Lyles M, Guermazi A, Bennell KL, Loeser RF. Effect of High-Intensity Strength Training on Knee Pain and Knee Joint Compressive Forces Among Adults With Knee Osteoarthritis: The START Randomized Clinical Trial. JAMA. 2021 Feb 16;325(7):646-657. doi: 10.1001/jama.2021.0411. PMID 33591346
- [Background] Dantas G, Sacco ICN, Dos Santos AF, Watari R, Matias AB, Serrao PRMS, Pott-Junior H, Salvini TF. Effects of a foot-ankle strengthening programme on clinical aspects and gait biomechanics in people with knee osteoarthritis: protocol for a randomised controlled trial. BMJ Open. 2020 Sep 25;10(9):e039279. doi: 10.1136/bmjopen-2020-039279. PMID 32978204
- [Background] Samuel AJ, Kanimozhi D. Outcome measures used in patient with knee osteoarthritis: With special importance on functional outcome measures. Int J Health Sci (Qassim). 2019 Jan-Feb;13(1):52-60. PMID 30842718
- [Background] Hashimoto T, Sakuraba K. Strength training for the intrinsic flexor muscles of the foot: effects on muscle strength, the foot arch, and dynamic parameters before and after the training. J Phys Ther Sci. 2014 Mar;26(3):373-6. doi: 10.1589/jpts.26.373. Epub 2014 Mar 25. PMID 24707086
- [Background] Kim I, Kim HA, Seo YI, Song YW, Hunter DJ, Jeong JY, Kim DH. Tibiofemoral osteoarthritis affects quality of life and function in elderly Koreans, with women more adversely affected than men. BMC Musculoskelet Disord. 2010 Jun 22;11:129. doi: 10.1186/1471-2474-11-129. PMID 20569450